CLINICAL TRIAL: NCT06895707
Title: Clinical Evaluation of BioFlx Crowns and Preformed Zirconia Crowns on Primary Second Molars: a Randomized Clinical Trial
Brief Title: Clinical Evaluation of BioFlx Crowns and Preformed Zirconia Crowns on Primary Second Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Fatimah alsuwaiyan, Resident, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPGRP/2024/822/1146/1065
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Clincal Evaluation of BioFlx Vs. Zirconia Crowns

STUDY DESIGN:
Masking Description: Data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Primary lower second molar (Experimental): one NuSmile® BioFlx crown will be placed on primary lower second molar.
  Interventions: Other: BioFlx crown
- Contralateral primary lower second molar (Active Comparator): one zirconia crown will be placed on the contralateral primary lower second molar.
  Interventions: Other: Zirconia crown

INTERVENTIONS:
Other: BioFlx crown — NuSmile® BioFlx crown (Group A) will be placed on primary lower second molar.
  Arms: Primary lower second molar
Other: Zirconia crown — Zirconia crown (Group B) will be placed on the contralateral primary lower second molar.
  Arms: Contralateral primary lower second molar

SUMMARY:
The goal of this clinical trial is to clinically evaluate the performance of BioFlx in comparison to preformed zirconia crowns in the restoration of primary second molars in pediatric patients.

The main questions it aims to answer are:

Is there a difference between BioFlx crowns (Group A) and one zirconia (Group B) in terms of crown retention (primary outcome)? Is there a difference between BioFlx crowns (Group A) and one zirconia (Group B) in modified gingival index, plaque index, occlusion, surface roughness, stain resistance, wear of opposing tooth, color match, anatomic form, marginal integrity and discoloration, proximal contact, and recurrent caries at the crown margins?

Researchers will compare the clinical performance of Bioflx crowns and zirconia crowns to determine if they are similar.

Participants:

* Participants will be asked to attend two appointments. During the first visit, a BioFlx crown will be placed on the primary lower second molar, and during the second visit, a zirconia crown will be placed on the contralateral primary lower second molar.
* Participants will be recalled and evaluated after 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-9 years old.
* American Society of Anesthesiologists Classification I or II status.
* Cooperative child.
* Obtained informed consent.
* Two primary lower second molars requiring full coverage restorations.
* Primary lower second molars in functional occlusion with the opposing tooth and have at least one contact area with an adjacent tooth.
* Primary lower second molars that can be adequately isolated.
* Pulptomized primary lower second molars.
* Primary lower second molars with multi-surface caries.

Exclusion Criteria:

* American Society of Anesthesiologists Classification higher or equal to three statuses.
* Informed consent is not obtained.
* Allergy to local anesthesia.
* Non-restorable primary lower second molars.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Crown retention | 3, 6, 12 months
  Evaluate whether the crown is present or absent 0= present
  1= absent

SECONDARY OUTCOMES:
Modified gingival index | 3, 6, 12 months
  0= normal
  1. mild inflammation
  2. moderate inflammation
  3. sever inflammation
Plaque index | 3, 6, 12 months
  Plaque index 0= no plaque
  1. film at gingival margin
  2. moderate accumulation
  3. abundance of plaque
Occlusion | 3, 6, 12 months
  0= clinically ideal with crown in harmony with occlusion
  1. clinically acceptable with crown occluding slightly high or low
  2. clinically unacceptable and crown needs to be replaced
Surface roughness | 3, 6, 12 months
  0= clinically ideal with smooth crown surface
  1. clinically acceptable with slight rough surface
  2. clinically unacceptable with crown fracture or pitting that require replacement
Stain resistance | 3, 6, 12 months
  0= no staining
  1. minor staining that can be polished
  2. noticeable staining that cannot be polished
Wear of opposing tooth | 3, 6, 12 months
  0= no wear
  1. mild wear
  2. severe wear
Color match | 3, 6, 12 months
  0= no color mismatch
  1. acceptable crown with color mismatch
  2. unacceptable crown with color mismatch
Anatomic form | 3, 6, 12 months
  0= clinically ideal
  1. clinically acceptable (slightly under/over contoured)
  2. clinically unacceptable (crown is missing or causing pain)
Marginal integrity and discoloration | 3, 6, 12 months
  0= clinically ideal
  1. clinically acceptable with slight discoloration
  2. clinically unacceptable with clear discoloration
Proximal contact | 3, 6, 12 months
  0= clinically ideal with acceptable resistance to the passage of floss
  1. clinically acceptable with tight or loose passage of floss
  2. clinically unacceptable with no contact with adjacent tooth
Recurrent caries | 3, 6, 12 months
  0= clinically ideal with no presence of recurrent caries
  1= clinically unacceptable with evidence of recurrent caries